CLINICAL TRIAL: NCT03693339
Title: An Open-label, Multicenter, Phase II Study of Capmatinib in Patients With Non-small Cell Lung Cancer Harboring MET Exon 14 Skipping Mutation
Brief Title: Capmatinib in Patients With Non-small Cell Lung Cancer Harboring cMET exon14 Skipping Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sang-We Kim, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STARTER_cMET
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Cancer; Lung Cancer Metastatic; MET Gene Mutation
MeSH Terms: conditions — Neoplasms | interventions — capmatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Capmatinib (Experimental): Capmatinib 400 mg twice oral administration and continuously dosing (28-day treatment schedule as one treatment cycle)
  Interventions: Drug: Capmatinib

INTERVENTIONS:
Drug: Capmatinib — Capmatinib 400 mg twice oral administration and continuously dosing (28-day treatment schedule as one treatment cycle)

SUMMARY:
This study is a phase II, single-arm, open label study under an umbrella trial for NSCLC. This clinical study is targeted for the patients who harbor exon 14 skipping mutation of MET and all patients will be treated with Capmatinib. The treatment period begins on Day 1 of Cycle 1 and 1 cycle consists of 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically or cytologically confirmed, unresectable stage IIIB/IV NSCLC that carries MET exon 14 skipping alteration by molecular testing, as per NGS and RT PCR.
* ECOG performance status of 0 to 2
* Male or female; ≥ 18
* Subjects with measurable lesion (using RECIST 1.1 criteria)
* Subjects must have archival tissue sample available, collected either at the time of diagnosis of NSCLC or any time since
* Patients who have progressed during or after 1st line or 2nd line therapy prior to the first dose of capmatinib. For patient who have received prior platinum containing adjuvant, neoadjuvant, or definitive chemoradiation for locally advanced disease, those treatments are regarded as 1st line if the progression has occurred < 12 months from last therapy.

Exclusion Criteria:

* Any major operation or irradiation within 4 weeks of baseline disease assessment
* Any clinically significant gastrointestinal abnormalities which may impair intake or absorption of the study drug
* Subjects with symptomatic central nervous system (CNS) metastases who are neurologically unstable or have required increasing doses of steroids within the 2 weeks prior to study entry to manage CNS symptoms
* Patients who have received more than 2 lines of prior systemic therapy, which include chemo, immune and targeted therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2018-10-30 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | At Week 6 then every 6 weeks up to Week 36.and then every 12 weeks until discharge, for an average of 13.8 months]
  ORR is a proportion of patients with a best overall response defined as complete response or partial response by RECIST1.1

SECONDARY OUTCOMES:
Duration of response | At Week 6 then every 6 weeks up to Week 36.and then every 12 weeks until discharge, for an average of 13.8 months
  DOR is calculated as the time from the date of the first document of complete remission (CR) or partial remission (PR) to the first documented preogressive disease (PD) or death due to any cause for patients with PR or CR.
Progression-free survival | At Week 6 then every 6 weeks up to Week 36.and then every 12 weeks until discharge, for an average of 13.8 months
  PFS is defined as time from the first dose of investigational products (IPs) to progression or death due to any cause.
  OS is defined as time from the first dose of IPs to death due to any cause.
Overall survival | At Week 6 then every 6 weeks up to Week 36.and then every 12 weeks until discharge, for an average of 13.8 months

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided